CLINICAL TRIAL: NCT02531854
Title: A Phase 2, Open-label, Randomized, Parallel Group, Controlled Study of Pemetrexed Maintenance With or Without ADXS11-001 Immunotherapy in Patients With Human Papillomavirus-Positive, Non-Squamous, Non-Small Cell Lung Carcinoma Following First-Line Induction Chemotherapy
Brief Title: A Study of Pemetrexed Maintenance With or Without ADXS11-001 Immunotherapy in Patients With Human Papillomavirus Positive (HPV+), NSCLC Following First-Line Induction Chemotherapy
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was withdrawn per sponsor decision
Sponsor: Advaxis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GBP-11-201
Record Dates: First submitted 2015-02-26; First posted 2015-08-25 (Estimated); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ADXS11-001 + Pemetrexed (Experimental)
  Interventions: Drug: ADXS11-001; Drug: Pemetrexed
- Pemetrexed Only (Active Comparator)
  Interventions: Drug: Pemetrexed

INTERVENTIONS:
Drug: ADXS11-001 — ADXS11-001 is a live attenuated Listeria monocytogenes (Lm) bacteria bioengineered to secrete an antigen-adjuvant fusion protein (tLLO¬HPV-E7) consisting of a truncated fragment of the listeriolysin O (tLLO) fused to the full length E7 peptide of HPV-16.
  Arms: ADXS11-001 + Pemetrexed
Drug: Pemetrexed — Chemotherapy

SUMMARY:
* Open label
* Enrollment in the order of confirmation of eligibility and HPV+ tumor status
* Prospective stratification based on 3 factors, epidermal growth factor receptor (EGFR) mutation status, performance status and first-line induction chemotherapy outcome;
* Randomization (2:1 ratio): (82 patients receiving the combination of pemetrexed plus ADXS11-001 vs. 42 patients receiving pemetrexed alone)
* Treatment Arm: Pemetrexed plus ADXS11-001 immunotherapy
* Control Arm: Pemetrexed only
* Positive control: pemetrexed chemotherapy

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients, ≥ 20 years of age
2. Patients with NSCLC
3. Patients whose disease has either responded or not progressed following 4-6 cycles of first-line induction chemotherapy.
4. Patients with documented/confirmed intra-tumor positivity for HPV
5. Patients with no major existing co-morbidities or medical conditions that will preclude administration of therapy, in the opinion of the Investigator
6. Patients with Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1
7. Patients will use contraception during the study
8. Patients with the ability to understand and give written informed consent for participation in this trial

Exclusion Criteria:

1. Women who are pregnant or breast feeding
2. Patients with histologically- or cytologically-confirmed squamous cell-classified NSCLC
3. Patients with disease progression following first-line induction chemotherapy
4. Patients with known active and uncontrolled central nervous system (CNS) or leptomeningeal metastases
5. Patients with an active second primary malignancy or history of another malignancy
6. Patients with inadequate recovery from an acute toxicity associated with any prior antineoplastic therapy, including ≥ Grade 2 neuropathy
7. Patients with inadequate recovery from any previous surgical procedure, or patients having undergone any major surgical procedure within 4 weeks prior to the start of study treatment
8. Patients with evidence of inadequate organ function as defined in protocol
9. Patients with a known allergy to both of the following antibiotics: ampicillin, trimethoprim-sulfamethoxazole
10. Patients with a known allergy to anti-emetic medications and/or non-steroidal anti-inflammatory drugs (e.g., ibuprofen, naproxen, celecoxib)
11. Patients with a history of severe hypersensitivity reaction to pemetrexed disodium (Alimta® or equivalent), or any of the excipients used in its formulation
12. Patients with a history of an autoimmune disorder requiring systemic treatment within the past 3 months, or a documented history of a clinically severe autoimmune disease or a syndrome that requires systemic steroid or immunosuppressive agents
13. Patients with a known immunodeficiency including patients: with HIV infection, who have undergone previous organ transplantation and require immunosuppressive therapy or long-term immunosuppressive therapy for any other reason
14. Patients with interstitial lung disease or active, non-infectious pneumonitis, active or prior documented inflammatory bowel diseases (e.g., Crohn's disease, ulcerative colitis)
15. Patients with an active infection requiring systemic therapy, prior to dosing with study drug
16. Patients with any other life-threatening illness, uncontrolled medical condition (e.g., elevated troponin or creatinine; uncontrolled diabetes), significant organ system dysfunction, or clinically significant laboratory abnormality, which in the opinion of the Investigator would either compromise the patient's safety or interfere with evaluation of the study treatment
17. Patients with a psychiatric disorder, substance abuse disorder, or altered mental status that would preclude understanding of the informed consent process and/or completion of the necessary study-related evaluations
18. Patients with a history of or current evidence of any condition, therapy, or laboratory abnormality that might: confound the results of the trial, interfere with the patient's participation in the trial, or suggest that participation in the trial is not in the best interest of the patient, in the opinion of the treating investigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-12 (Estimated); Primary Completion 2019-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Number of study participants with objective tumor response as assessed by Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1 and Immune-Related Response Evaluation Criteria in Solid Tumors (irRECIST) | 2 years
Number of study participants with progression free survival as assessed by Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1 and Immune-Related Response Evaluation Criteria in Solid Tumors (irRECIST) | 2 years

SECONDARY OUTCOMES:
Distribution of overall response rate (ORR) as assessed by RECIST v1.1 and irRECIST | 2 years
Distribution of duration of response (DR) as assessed by RECIST v1.1 and irRECIST | 2 years
Distribution of disease stabilization (SD) as assessed by RECIST v1.1 and irRECIST | 2 years
Distribution of overall survival (OS) as assessed by RECIST v1.1 and irRECIST | 2 years
Frequency and severity of treatment related adverse events (AEs) as assessed by Common Terminology Criteria for Adverse Events (CTCAE) v4.03 for study participants on the combination arm | 2 years